CLINICAL TRIAL: NCT07141862
Title: Fertility Preservation in Children With Neuroblastoma or Ewing's Sarcoma: Detection of Residual Disease by a Sensitive Method
Brief Title: Fertility Preservation in Children With Solid Tumors: Detection of Residual Disease by a Sensitive Method
Acronym: PREFERPUBER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2025_BRUGNON_PREFERPUBER
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma; Ewing Sarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Detection of MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues using RT-qPCR: First, the detection of minimal residual disease of neuroblastoma and Ewing sarcoma will be performed on an in vitro model that mimics the metastatic dissemination of these two solid tumors. Ovarian and testicular tissues will be contaminated with increasing quantities of tumor cells (0, 5, 10, 20, and 100 tumor cells) from neuroblastoma (IMR-32) and Ewing sarcoma (RD-ES). Then, the detection of MRD will be carried out on ovarian and testicular tissues from prepubertal patients diagnosed and treated for neuroblastoma and Ewing sarcoma during infancy.
  To detect this MRD in both models, the investigators will perform RNA extraction using TRIzol reagent, followed by reverse transcription and RT-qPCR to detect the specific tumor genes: PHOX2B for neuroblastoma and EWSR1-FLI1 for Ewing sarcoma.
  Interventions: Diagnostic Test: RT-qPCR
- Detection of MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues using ddPCR.: First, the detection of MRD of neuroblastoma and Ewing sarcoma will be performed on an in vitro model that mimics the metastatic dissemination of these two solid tumors. Ovarian and testicular tissues will be contaminated with increasing quantities of tumor cells (0, 5, 10, 20, and 100 tumor cells) from neuroblastoma (IMR-32) and Ewing sarcoma (RD-ES). Then, the detection of MRD will be carried out on ovarian and testicular tissues from prepubertal patients diagnosed and treated for neuroblastoma and Ewing sarcoma during infancy.
  To detect this MRD in both models, the investigators will perform RNA extraction using TRIzol reagent, followed by reverse transcription and ddPCR to detect the specific tumor genes: PHOX2B for neuroblastoma and EWSR1-FLI1 for Ewing sarcoma.
  Interventions: Diagnostic Test: ddPCR

INTERVENTIONS:
Diagnostic Test: RT-qPCR — Detection of MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues using RT-qPCR
  Groups: Detection of MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues using RT-qPCR
Diagnostic Test: ddPCR — Detection of MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues using ddPCR
  Groups: Detection of MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues using ddPCR.

SUMMARY:
In prepubertal patients, cryopreservation of ovarian or testicular tissue is currently the only available method for fertility preservation prior to gonadotoxic cancer treatments. However, this approach carries the risk of reintroducing malignant cells upon autotransplantation, particularly in cases of metastatic cancers such as neuroblastoma and Ewing sarcoma. Therefore, it is crucial to employ highly sensitive techniques to detect minimal residual disease (MRD) in preserved gonadal tissues.

This study aims to identify the most effective detection method by comparing the sensitivity and specificity of reverse transcription quantitative PCR (RT-qPCR) and droplet digital PCR (ddPCR) in identifying MRD of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues from patients treated for these malignancies during infancy.

DETAILED DESCRIPTION:
Ovarian and testicular cryopreservation is the only option to preserve the fertility of children diagnosed with cancer. Cancer treatments such as chemotherapy and radiotherapy can lead to gonadal toxicity. However, there is a risk of reintroducing tumor cells when the germinal tissue is reused. This is known as residual disease. This risk is higher in the case of metastatic cancers such as neuroblastoma and Ewing sarcoma. These two solid tumors are associated with a high risk of relapse and disease progression after treatment. Neuroblastoma is the most common extracranial solid tumor in children. One characteristic of this neuroendocrine tumor is its high frequency of metastatic disease. Several cases of metastasis have been reported in ovarian and testicular tissues.

Regarding Ewing sarcoma, it is the second most common bone cancer in children. Approximately 27% of patients show evidence of metastasis at diagnosis; these circulating tumor cells can reach the germinal tissues.

Several detection methods are available for these two solid tumors, such as histopathological analysis with hematoxylin-eosin staining, and immunohistochemistry targeting cellular markers with fluorescent antibodies. However, the main limitation of these two methods is their low sensitivity for detecting only a few tumor cells. That is why RT-qPCR and ddPCR, which have high detection sensitivity, have been developed. These two molecular methods are currently used for the detection of residual disease in leukemia and lymphoma. However, no studies have investigated the detection of residual disease of neuroblastoma and Ewing sarcoma by ddPCR in ovarian and testicular tissues.

Therefore, the goal of this study is to validate the detection of residual disease of neuroblastoma and Ewing sarcoma by ddPCR in ovarian and testicular tissues. In addition, the second goal is to evaluate the specificity and sensitivity of residual disease detection for these two solid tumors in ovarian and testicular tissues using RT-qPCR and ddPCR.

First, an in vitro model has been developed to mimic the metastatic dissemination of neuroblastoma and Ewing sarcoma in germinal tissues. To do this, two tumor cell lines will be used: IMR-32 for neuroblastoma and RD-ES for Ewing sarcoma. Then, 10 ovarian tissues and 10 testicular tissues will be contaminated with increasing quantities of neuroblastoma tumor cells: 5, 10, 20, and 100 tumor cells. The same procedure will be applied in the case of Ewing sarcoma. Ovarian tissues are derived from women of any age diagnosed with a benign cyst requiring laparoscopy. Testicular tissues are derived from men of any age diagnosed with non-obstructive azoospermia. These ovarian and testicular models have been validated by our team through preliminary work. These models are as close as possible to prepubertal tissues with immature gametes. Next, the investigators will perform RNA extraction with TRIzol reagent, followed by reverse transcription to generate complementary DNA (cDNA) and RT-qPCR and ddPCR to detect the specific tumor genes: PHOX2B for neuroblastoma and EWSR1-FLI1 for Ewing sarcoma.

Residual disease detection will be conducted on ovarian and testicular tissues collected from prepubertal patients diagnosed and treated for neuroblastoma or Ewing sarcoma during infancy. These patients underwent germinal tissue cryopreservation as a fertility preservation strategy following their cancer diagnosis.

Total RNA will be extracted from the cryopreserved tissues using TRIzol reagent. Subsequently, reverse transcription will be performed. The presence or absence of tumor-specific transcripts will be assessed using both reverse transcription quantitative PCR (RT-qPCR) and droplet digital PCR (ddPCR). Specifically, the neuroblastoma-associated PHOX2B gene and the Ewing sarcoma-specific EWSR1-FLI1 fusion transcript will be targeted.

By comparing the sensitivity and specificity of RT-qPCR and ddPCR for detecting minimal residual disease in these tissues, this study aims to determine the most effective and reliable protocol for identifying residual tumor cells. The findings will support the safe future use of cryopreserved ovarian and testicular tissues in fertility restoration for pediatric cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age diagnosed with a benign cyst requiring laparoscopy may be included.
* Men of any age diagnosed with a non-obstructive azoospermia may be included.
* Prepubertal girls and boys diagnosed with neuroblastoma or Ewing sarcoma during infancy may be included.
* Capable of providing written informed consent to participate in the research study
* Affiliated with a social welfare service.
* For prepubertal patients, written informed consent to participate in the research study must be provided by their parents or legal guardians.

Exclusion Criteria:

* None

Ages: 2 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: Residual disease detection will be conducted on ovarian and testicular tissues collected from prepubertal patients diagnosed and treated for neuroblastoma or Ewing sarcoma during infancy
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of residual disease detection of neuroblastoma and Ewing sarcoma by ddPCR in ovarian and testicular tissues. | From 02-2025 to 02-2026 for analysis of neuroblastoma; from 02-2026 to 12-2027 for analysis of Ewing sarcoma.
  Detection of the copy number of specific tumor genes: PHOX2B for neuroblastoma and EWSR1-FLI1 for Ewing sarcoma in ovarian and testicular tissues using ddPCR. Residual disease will be detected in ovarian and testicular tissues contaminated with increasing quantities of tumor cells (0, 5, 10, 20, and 100 tumor cells) from neuroblastoma (IMR-32) and Ewing sarcoma (RD-ES), as well as in ovarian and testicular tissues from prepubertal patients diagnosed and treated for neuroblastoma and Ewing sarcoma during infancy.

SECONDARY OUTCOMES:
Evaluation of the specificity and sensitivity of RT-qPCR and ddPCR for detecting residual disease of neuroblastoma and Ewing sarcoma in ovarian and testicular tissues. | From 02-2025 to 02-2026 for analysis of neuroblastoma; from 02-2026 to 12-2027 for analysis of Ewing sarcoma.
  Detection of the copy number of specific tumor genes: PHOX2B for neuroblastoma and EWSR1-FLI1 for Ewing sarcoma in ovarian and testicular tissues using RT-qPCR and ddPCR. Residual disease will be detected in ovarian and testicular tissues contaminated with increasing quantities of tumor cells (0, 5, 10, 20, and 100 tumor cells) from neuroblastoma (IMR-32) and Ewing sarcoma (RD-ES), as well as in ovarian and testicular tissues from prepubertal patients diagnosed and treated for neuroblastoma and Ewing sarcoma during infancy. The sensitivity and specificity of each detection method will then be compared.
Evaluation of the impact of ovarian tissue freezing protocols on RNA Quantity and Purity | From 02-2025 to 02-2026 for analysis of neuroblastoma; from 02-2026 to 12-2027 for analysis of Ewing sarcoma
  Two ovarian tissue freezing protocols will be tested. Half of the ovarian tissues contaminated by neuroblastoma tumor cells (IMR-32) will be frozen and thawed using the protocol describe by Gosden in 1994, and the other half using the protocol developed by Schubert in 2005. RNA quantity and purity, including protein and chemical contamination will be compared between the two protocols.
  The same analysis will be performed on ovarian tissues contaminated with Ewing sarcoma tumor cells (RD-ES).

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, MD, PhD, HDR, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University hospital, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: Undecided